CLINICAL TRIAL: NCT05524506
Title: PROgnostic Value of MicroParticles and Markers of Hemostasis in TIA and Ischemic Stroke
Acronym: PROMPTS
Status: Completed | Type: Observational
Sponsor: Karolinska Institutet (Other)
Collaborators: Danderyd Hospital (Other); Stockholm South General Hospital (Other)
Responsible Party: Principal Investigator, Ann Charlotte Laska, Associate professor, Karolinska Institutet
Other Study IDs: KIDS-IM-LL-2016-01
Record Dates: First submitted 2020-09-23; First posted 2022-09-01 (Actual); Last update posted 2022-09-01 (Actual); Status verified 2022-08

CONDITIONS: Brain Ischemia; Cerebral Ischemia; Extracellular Vesicles; Hemostasis; Prognosis
Keywords: Ischemic stroke; TIA; Microparticles; Markers of hemostasis; Stroke etiology
MeSH Terms: conditions — Brain Ischemia; Ischemic Stroke

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — Platelet-poor plasma (citrated and EDTA)
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
The purpose is to investigate if different microparticles and markers of hemostasis predict outcome after TIA or ischemic stroke and to study the association between these variables and stroke subtype or etiology.

DETAILED DESCRIPTION:
1. Introduction Within a previous study ('PROPPSTOPP') a cohort of 249 patients with ischemic stroke (IS) or TIA was established in Stockholm between 2007 and 2009. The original aims were twofold: 1) to look for occult atrial fibrillation (completed, NTC01160406) and 2) to investigate microparticle levels and markers of hemostasis in the acute phase and one month after symptoms. Blood samples were taken on both occasions. Patients were found to have higher microparticle levels and increased thrombin generation in plasma both acutely and at one month as compared to healthy controls.

   This follow-up study will investigate the prognostic ability of microparticles (primary variables) and markers of hemostasis (secondary variables) to predict outcome as documented in hospital records and Swedish registers. The association between microparticles/coagulation markers and stroke subtype/etiology will also be investigated.
2. Variables

   2.1 Microparticles

   Microparticles are membrane vesicles (0.1-1.0 µm) released from cells at activation or apoptosis. They carry surface markers from the releasing cell. Microparticles are of interest as biomarkers for activation of cells in the circulation, e g platelets, endothelial cells or leukocytes. They may have pro-coagulant properties. For this study the following microparticles and surface markers have been analyzed:
   * Total number of microparticles (MP's)
   * Number of MP's exposing phosphatidylserine (PS) (pro-coagulant property)
   * Number of MP's of any type exposing tissue factor (TF), with or without simultaneous exposure of PS (pro-coagulant properties, activation of monocytes/endothelium)
   * Number of platelet microparticles (PMP's), identified by surface exposure of GPαIIb (CD41), with or without simultaneous exposure of PS (platelet activation)
   * Number of PMP's exposing P-selectin with or without simultaneous exposure of PS (platelet activation)
   * Number of PMP's exposing TF with or without simultaneous exposure of PS (pro-coagulant properties)

   2.2 Markers of hemostasis

   Different variables of importance for coagulation, platelet activation, fibrinolysis and inflammation were measured in the original study, namely:
   * Prothrombin fragment F1+2
   * Thrombin generation by Calibrated Automated Thrombin generation (CAT)
   * Microparticle-pellet induced thrombin generation
3. Outcome

   3.1 Primary outcome

   The primary outcome is new ischemic events, i e fatal or non-fatal recurrent ischemic stroke, myocardial infarction or ischemic cardiovascular death in the time frame 2007-2014. Diagnoses will be retrieved from the following sources:
   * The Swedish Register for Cause of death
   * The Swedish Register of in-house hospital care
   * Medical records at recruiting hospitals.

   3.2 Secondary outcome

   Secondary outcomes are recurrent ischemic stroke respectively all-cause mortalitý as documented in the sources above.
4. Statistical Methods

The statistical analysis of the prospective cohort study will be performed in steps:

1. Descriptive statistics comparing averages/medians of the above variables for patients with and without outcome.
2. For variables with p-values < 0.2 in step 1: univariate event-free survival Kaplan-Meyer curves by variable median split. Probability calculations of differences by log-rank test.
3. Multivariate analysis by Cox regression analysis including the most significant variables in step 2 and established cardiovascular risk factors.

ELIGIBILITY:
Cohort established in NTC01160406

Inclusion Criteria:

* acute ischemic stroke or TIA less than 2 weeks before enrollment
* ability to understand study instructions both verbal and written
* ability to handle handheld ECG

Exclusion Criteria:

* known atrial fibrillation
* hemorrhagic stroke at time of enrollment
* limited compliance
* pacemaker

Min Age: 45 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Patients from two hospital stroke units in Stockholm having suffered ischemic stroke or TIA 2007-2009 without known atrial fibrillation and able to handle handheld ECG-recorder.
Sampling Method: Non-Probability Sample
Enrollment: 249 (Actual)
Dates: Start 2007-06 (Actual); Primary Completion 2014-12 (Actual); Study Completion 2021-06-30 (Actual)

PRIMARY OUTCOMES:
Fatal or non-fatal ischemic stroke or myocardial infarction. | 2007-2014
  New fatal or non-fatal ischemic stroke after the initial ischemic stroke or TIA leading to recruitment. Outcome events and time of events are extracted from national registries ('Patientregistret', 'Dödsorsaksregistret') and hospital records.

SECONDARY OUTCOMES:
Recurrent ischemic stroke | 2007-2014
  Recurrent ischemic stroke (fatal or non-fatal) after initial ischemic stroke or TIA leading to recruitment. Outcome events and time of events are extracted from national registries ('Patientregistret') and hospital records.
All-cause mortality | 2007-2014
  All cause mortality after initial ischemic stroke or TIA leading to recruitment. Outcome events and time of events are extracted from national registry ('Dödsorsaksregistret').

CONTACTS AND LOCATIONS:
Overall Officials: Mårten Rosenqvist, Prof, Principal Investigator — Karolinska Institutet
Locations (1):
- Karolinska Institutet, Daderyd Hospital, Stockholm, Sweden

IPD SHARING:
Plan to Share IPD: No
Not intended at present.

REFERENCES:
- [Background] Lundstrom A, Mobarrez F, Rooth E, Thalin C, von Arbin M, Henriksson P, Gigante B, Laska AC, Wallen H. Prognostic Value of Circulating Microvesicle Subpopulations in Ischemic Stroke and TIA. Transl Stroke Res. 2020 Aug;11(4):708-719. doi: 10.1007/s12975-019-00777-w. Epub 2020 Jan 25. PMID 31983048
- [Background] Lundstrom A, Anggardh-Rooth E, Mobarrez F, Thalin C, Gigante B, Laska AC, Wallen H. High Thrombin Generation after Acute Ischemic Stroke or Transient Ischemic Attack Is Associated with a Reduced Risk of Recurrence: An Observational Cohort Study. Thromb Haemost. 2021 May;121(5):584-593. doi: 10.1055/s-0040-1721146. Epub 2020 Dec 12. PMID 33314013